CLINICAL TRIAL: NCT05904145
Title: Pregnancy Risk, Infant Surveillance, and Measurement Alliance (PRiSMA) Maternal and Newborn Health (MNH) Study: A Multi-center, Prospective Cohort Study of Maternal, Newborn, and Infant Health
Brief Title: PRISMA Maternal and Newborn Health Study
Acronym: PRiSMA-MNH
Status: Recruiting | Type: Observational
Sponsor: George Washington University (Other)
Collaborators: Kenya Medical Research Institute (Other); University of North Carolina, Chapel Hill (Other); Kintampo Health Research Centre, Ghana (Other); Aga Khan University (Other); Christian Medical College, Vellore, India (Other); Centres for Disease Control and Prevention, Kenya. (Other); Vital Pakistan Trust (Other)
Responsible Party: Principal Investigator, Emily Smith, Princiapl Investigator, George Washington University
Other Study IDs: PRiSMA-MNH 2022
Record Dates: First submitted 2022-10-14; First posted 2023-06-15 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Pregnancy, High Risk
Keywords: Antenatal Care (ANC); Postnatal Care (PNC); Maternal Newborn Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Access to quality antenatal care (ANC) and postnatal care (PNC), including maternal, newborn, and infant services, is integral to reducing adverse pregnancy-related health outcomes and promoting positive birth experiences. The World Health Organization (WHO) recommends a total of eight ANC visits for pregnant women. However, the ANC coverage rate remains considerably lower among more vulnerable populations, and the quality of care that women receive is inconsistent, often poor, and frequently fails to detect risks in a timely fashion or adequately prepare women for the birth process. While rates of facility-based delivery are on the rise worldwide, disparities persist and the quality of care across facilities remains uneven. Even less information is available on PNC, where services beyond routine immunizations may not be widely available, especially in resource-poor regions.

Additionally, limited evidence exists on innovative service delivery approaches and how to effectively scale tested maternal and newborn health (MNH) interventions. This coupled with the fragmented datasets from smaller studies limit our ability to advocate for policy change.

The Pregnancy Risk Stratification Innovation and Measurement Alliance (PRiSMA) is implementing a harmonized open cohort study that seeks to evaluate pregnancy risk factors and their associations with adverse pregnancy outcomes, including stillbirth, neonatal mortality and morbidity, and maternal mortality and severe morbidity. The goals are to develop a harmonized data set to improve understanding of pregnancy risk factors, vulnerabilities, and morbidity and mortality and to estimate the burden of these risk factors and outcomes in LMICs. Ultimately, these data will inform development of innovative strategies to optimize pregnancy outcomes for mothers and their newborns.

ELIGIBILITY:
A woman who meets the following inclusion criteria during screening may be enrolled:

* Lives within the study catchment area;
* Meets minimum age requirement in study site country:

  * Ghana: 15 years of age;
  * Kenya: 18 years of age or those who meet the criteria of emancipated minors;
  * Pakistan: 15 years of age or those who meet the criteria of emancipated minors;
  * Zambia: 15 years of age;
  * India: 18 years of age
* Intrauterine pregnancy <20 weeks gestation verified via ultrasound;
* Provides informed consent.

A woman who meets the following exclusion criteria during screening may NOT be enrolled:

* Nonviable (e.g. ectopic or molar) pregnancy;
* Plans to relocate outside of the study catchment area during pregnancy and/or postpartum.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The investigators will identify, screen, and enroll pregnant participants through pregnancy surveillance systems, with a goal of identifying pregnancies prior to 20 weeks of pregnancy. Pregnant women will be assessed at <20, 20, 28, 32, and 36 weeks gestation, at labor and delivery, and at 3 days and 1, 4, 6, 26, and 52 weeks postpartum. Infants will similarly be assessed at 3 days and 1, 4, 6, 26, and 52 weeks of age.
Sampling Method: Non-Probability Sample
Enrollment: 267897 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Maternal Mortality | Assessed from time of pregnancy identification (on average, 10-20 weeks gestational age), through delivery or termination of pregnancy, and then 42 days postpartum
  Death from any cause related to or aggravated by pregnancy or its management (excluding accidental or incidental causes) during pregnancy and childbirth or within 42 days of termination of pregnancy, irrespective of the duration and site of the pregnancy.
Composite Severe Maternal Outcomes | Assessed through 12 months postpartum
  Composite outcome of maternal deaths + near-miss cases + potentially life-threatening complications + critical intervention.
Maternal Anemia | Assessed from time of pregnancy identification (on average, 10-20 weeks gestational age) through 6 months postpartum
  Low hemoglobin levels throughout pregnancy and labor and delivery, classified as mild (10-10.9 g/dL), moderate (7-9.9 g/dL), or severe (<7 g/dL). Low hemoglobin levels in the postpartum period, classified as mild (11-11.9 g/dL), moderate (8-10.9 g/dL), or severe (<8 g/dL).
Stillbirth | Assessed at delivery
  Delivery of a fetus showing no signs of life, as indicated by absence of breathing, heartbeat, pulsation of the umbilical cord, or definite movements of voluntary muscles. The primary definition for the study is death prior to delivery of a fetus at >=20 weeks of gestation (or >350 g weight, if gestational age is unavailable). Additionally, we will analyze time-specific definitions: Early stillbirth (20-27 weeks), Late stillbirth (28-36 weeks), Term stillbirth (>=37 weeks), and WHO stillbirth (>=28 weeks).
Neonatal Mortality | Assessed delivery to 28 days of life
  Death of a live-born baby during the first 28 days of life from any cause.
Preterm Birth | Assessed at delivery
  Delivery prior to 37 completed weeks of gestation of a birth (live or stillbirth). Further classified as extremely preterm (<28 weeks), very preterm (28-32 weeks), and moderate to late preterm (32-37 weeks). For these, gestational age at birth will be determined by the best obstetric estimate: last menstrual period, Ultrasound (method to be determined), and ACOG algorithm.
Low Birth Weight | Assessed at delivery or within 72 hours for home births
  Defined as birth weight <2500 g and very low birth weight <1500 g.
Small-for-Gestational-Age (SGA) | Assessed at delivery
  Combined gestational age information and birthweight will be used to further categorize into: preterm-SGA, preterm-AGA, term-SGA, term-AGA.

SECONDARY OUTCOMES:
Late Maternal Mortality | Assessed from 42 days postpartum up to one year
Preeclampsia | Assessed from time of pregnancy identification (on average, 10-20 weeks gestational age) through 42 days postpartum
Preterm Birth Indication | Assessed at delivery
Preterm Premature Rupture of Membranes (PPROM) | Assessed at <37 weeks of gestation
Gestational Hypertension | : Assessed from 20 weeks gestational age through delivery
Postpartum Hypertension | Assessed at delivery or time of pregnancy to 1 year postpartum
Gestational Diabetes | Assessed between 24 and 28 weeks gestation
Perinatal Depression, as measured using the Edinburgh Postnatal Depression Scale | Assessed at 20 and 32 weeks gestation and 6 weeks postpartum
  The minimum value is 0 and the maximum value is 30. Higher scores indicate that more severe depression may be present.
Maternal Infection and Sepsis | Assessed from time of pregnancy identification (on average, 10-20 weeks gestational age) through 42 days postpartum
Fetal Death | Assessed from time of pregnancy identification (on average, 10-20 weeks gestational age) up until delivery
Cause of Neonatal Death | Assessed at <28 days of life
Cause of Stillbirth | : Assessed from 20 weeks gestational age through time of delivery
Timing of Stillbirth | : Assessed from 20 weeks gestational age through time of delivery
Timing of neonatal mortality | Assessed from delivery to 28 days of life
Infant Mortality | Assessed from delivery to 1 year of life
Hyperbilirubinemia | Assessed at birth, 3 days, and 7 days of age
Neonatal Sepsis | Assessed at delivery through 28 days
Possible Severe Bacterial Infection | Assessed from delivery to 59 days
Postnatal Weight Trajectory | Assessed collected at birth, 3 days, 7 days, and 28 days
Infant Growth | Assessed at birth, 4 weeks, 6 weeks, 6 months, 26 months, and 52 months

CONTACTS AND LOCATIONS:
Locations (5):
- Kintampo Health Research Centre, Kintampo, Ghana
- Christian Medical College (CMC) Vellore, Vellore, India
- Kenya Medical Research Institute-Center for Global Health Research, Kisumu, Kenya
- Aga Khan University, Karachi, Pakistan
- University of North Carolina-Global Projects Zambia, Lusaka, Zambia

REFERENCES:
- [Derived] Pregnancy Risk, Infant Surveillance, and Measurement Alliance (PRISMA) Investigators. Pregnancy Risk, Infant Surveillance, and Measurement Alliance (PRISMA) Maternal and Newborn Health Study: protocol for a multisite, prospective, open cohort study of pregnancy and postpartum health outcomes in South Asia and sub-Saharan Africa. BMJ Open. 2026 Jan 20;16(1):e104512. doi: 10.1136/bmjopen-2025-104512. PMID 41558748
- [Derived] Smith ER, Hoodbhoy Z, Hotwani A, Jehan F, Khan A, Nisar I, Yazdani N, Benjamin SJ, Cherian AG, Mohan VR, Varghese S, Vijayalekshmi B, Wylie BJ, Chatterjee L, Dang A, Venketeshwar R, Baumann SG, Mores C, Pan Q, Sudfeld CR, Akelo V, Mwebia WK, Otieno K, Ouma G, Owuor H, Were J, Adu-Gyasi D, Agyemang V, Newton S, Tawiah C, Jadaun AS, Mazumder S, Sharma N, Ugwu LG, Benneh-Akwasi Kuma A, Freeman B, Kasaro MP, Mbewe FM, Mwape H, Resop RS, Spelke MB, Asante KP; Redefining Maternal Anemia in Pregnancy and Postpartum (ReMAPP) Study Investigators. Protocol for the Redefining Maternal Anemia in Pregnancy and Postpartum (ReMAPP) study: A multisite, international, population-based cohort study to establish global hemoglobin thresholds for maternal anemia. PLoS One. 2025 Jul 28;20(7):e0321943. doi: 10.1371/journal.pone.0321943. eCollection 2025. PMID 40720446
- [Derived] Naz S, Jaffar A, Yazdani N, Kashif M, Hussain Z, Khan U, Farooq F, Nisar MI, Jehan F, Smith E, Hoodbhoy Z. Cohort profile: the Pregnancy Risk Infant Surveillance and Measurement Alliance (PRISMA) - Pakistan. BMJ Open. 2023 Dec 10;13(12):e078222. doi: 10.1136/bmjopen-2023-078222. PMID 38072494